CLINICAL TRIAL: NCT06288815
Title: Comparison Efficacy of Oral Fluid Versus Intravenous Fluid Replacement in Postoperative Primary Total Knee Arthroplasty : A Randomized Controlled Trial.
Brief Title: Oral Fluid vs IV Fluid After Primary TKA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Yot Tanariyakul, Principle investigator, Thammasat University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUH oral fluid TKA
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee; Total Knee Arthroplasty; Oral Fluid Replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral fluid (Experimental): * NPO (8hr for food, 2hr for water)
  * Intraoperative IV fluid at least 1 liter
  * Post operative (Off IV fluid, allow oral fluid as protocol at least 24hr)
  Interventions: Dietary Supplement: Oral fluid
- IV fluid (Active Comparator): * NPO (8hr for food, 2hr for water)
  * Intraoperative IV fluid at least 1 liter
  * Post operative (IV fluid as protocol at least 24hr, allow oral fluid as usual)
  Interventions: Dietary Supplement: IV fluid

INTERVENTIONS:
Dietary Supplement: Oral fluid — Postoperation
  * Off IV fluid immediately postoperative
  * Allow patients drink oral fluid as protocol for 24hr
  Arms: Oral fluid
Dietary Supplement: IV fluid — Postoperation
  * IV fluid replacement as protocol for 24hr
  * Allow patients drink oral fluid as usual
  Arms: IV fluid

SUMMARY:
The goal of this study is to compared efficacy of oral fluid and intravenous fluid after primary unilateral total knee arthroplasty.

The main question it aims to answer is:

Does oral fluid replacement after primary unilateral total knee arthroplasty provide a patient recover faster than intravenous fluids replacement?

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85 years old
* ASA I, II
* Primary osteoarthritis

Exclusion Criteria:

* Diuretics use
* Morbid obesity
* Previous knee surgery
* Cannot undergo spinal anesthesia

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Time to stand and walk | Postoperative day 1
  Stand and walk with walker

SECONDARY OUTCOMES:
Time up and go | 24 and 48 hours
  Record time since stand up and walk 3 meters, or 10 feet away, on the floor
Incidence of oliguria | Postoperative day 1,2
  Urine output < 0.5ml/kg/hr
Incidence of nausea/vomiting | Postoperative day 1,2
  record symptom of nausea and vomiting
Urine specific gravity | Postoperative day 1
  Urine specific gravity every 4 hours
the levels of certain electrolytes | Postoperative day 1,2
  Blood chemistry
the levels of creatinine | Postoperative day 1,2
  Blood chemistry
the levels of blood urea nitrogen (BUN). | Postoperative day 1,2
  Blood chemistry
Complications | Until postoperative 3months
  Pulmonary edema, heart failure, acute kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jennings JM, Mejia M, Williams MA, Johnson RM, Yang CC, Dennis DA. The James A. Rand Young Investigator's Award: Traditional Intravenous Fluid vs. Oral Fluid Administration in Primary Total Knee Arthroplasty: A Randomized Trial. J Arthroplasty. 2020 Jun;35(6S):S3-S9. doi: 10.1016/j.arth.2020.01.029. Epub 2020 Jan 22. PMID 32037213